CLINICAL TRIAL: NCT02815995
Title: A Phase II Multi-Arm Study to Test the Efficacy of Immunotherapeutic Agents in Multiple Sarcoma Subtypes
Brief Title: Multi-Arm Study to Test the Efficacy of Immunotherapeutic Agents in Multiple Sarcoma Subtypes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-1071; NCI-2016-01178 (Other: NCI-CTRP Clinical Trials Reporting Registry)
Record Dates: First submitted 2016-06-16; First posted 2016-06-28 (Estimated); Results first posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-02

CONDITIONS: Advanced and/or Metastatic Sarcoma
Keywords: Malignant neoplasms of bone and articular cartilage; Multiple sarcoma subtypes; Advanced and/or metastatic sarcoma; Adipocytic tumors; Vascular tumors; Leiomyosarcoma; Angiosarcoma; Epithelioid hemangioendothelioma; Undifferentiated pleomorphic sarcoma; Synovial sarcoma; Osteosarcoma; Other sarcoma histologies; Durvalumab; Tremelimumab
MeSH Terms: conditions — Vascular Neoplasms; Leiomyosarcoma; Hemangiosarcoma; Hemangioendothelioma, Epithelioid; Histiocytoma, Malignant Fibrous; Sarcoma, Synovial; Osteosarcoma | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Adipocytic Tumors Group (Experimental): Adipocytic Tumors Group consists of well-diff/de-differentiated, pleomorphic and myxoid LPS.
  Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Vascular Tumors Group (Experimental): Vascular Tumors Group consists of leiomyosarcomas, angiosarcomas, epithelioid hemangioendotheliomas, and hemangiopericytomas.
  Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by Durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Undifferentiated Pleomorphic Sarcoma Group (Experimental): Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by Durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Synovial Sarcoma Group (Experimental): Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which Durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Osteosarcoma Group (Experimental): Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which Durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab
- Other Sarcomas Group (Experimental): Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which Durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — Age group ≥ 18: Durvalumab 1500 mg by vein every 4 weeks for 4 cycles. After Week 16, participant may continue to receive durvalumab alone by vein for an additional 32 weeks (8 doses).
Drug: Tremelimumab — Age group ≥ 18: Tremelimumab 75 mg every 4 weeks for 4 cycles.

SUMMARY:
The goal of this clinical research study is to learn if the combination of durvalumab and tremelimumab can help to control sarcoma. The safety of this drug combination will also be studied.

This is an investigational study. Durvalumab and tremelimumab are not FDA approved or commercially available. They are currently being used for research purposes only. The study doctor can explain how the study drugs are designed to work.

Up to 150 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Study Drug Administration:

If you are found to be eligible to take part in this study, you will receive tremelimumab and durvalumab by vein, over about 1 hour each, every 4 weeks for up to 16 weeks (4 doses). After Week 16, you may continue to receive durvalumab alone by vein over about 1 hour for an additional 32 weeks (8 doses).

If you have a side effect related to the combination of durvalumab and tremelimumab during the first 16 weeks of the study, you may be able to switch over to receive durvalumab alone sooner than expected. This will be discussed with you.

Study Visits:

On Day 1 of Week 0:

* You will have a physical exam.
* You will have 3 EKGs in a row.
* Blood (about 1 tablespoon) and urine will be collected for routine tests. If you can become pregnant, part of this routine blood and urine sample will be used for a pregnancy test.
* Blood (about 2½ tablespoons) will be drawn for biomarker and genetic testing. Biomarkers are found in the blood and may be related to your reaction to the study drug. The type of genetic testing in this study will be performed to learn how your DNA (genetic material) may change how you respond to the study drugs.

On Day 1 of Weeks 2 and 6, blood (about 3½ tablespoons) will be drawn for routine, genetic, and biomarker testing.

On Day 1 of Week 4 and then every 4 weeks after that (Weeks 8, 12, 16, and so on) until Week 44:

* You will have a physical exam.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* You will have imaging scans. You will not have these scans at Weeks 16 and 24.

On Day 1 of Weeks 10 and 14, blood (about 1 tablespoon) will be drawn for routine tests.

Length of Study:

You may receive up to 4 doses of durvalumab in combination with tremelimumab and up to an additional 8 doses of durvalumab alone. You will no longer be able to take the study drug(s) if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

If you complete 12 months of therapy but the disease appears to get worse, you may be able to re-start treatment. The study doctor will discuss this with you.

It is expected that your participation in this study may last up to 15 months. Your participation on the study will be over after the follow-up visits.

End-of-Treatment Visit:

As soon as possible after your last dose of study drug(s):

* You will have a physical exam.
* You will have an MRI, CT, or PET/CT scan.
* Blood (about 1 tablespoon) and urine will be collected for routine tests.
* Blood (about 1 tablespoon) will be drawn for biomarker and genetic testing.

Follow-Up Visit:

About 30 days after your last dose of study drug(s):

You will have a physical exam. Blood (about 1 tablespoon) will be drawn for routine tests.

Long-Term Follow-Up

Every 3 months:

* You will have an MRI, CT, or PET/CT scan.
* You may be called to learn how you are doing and if you have started any anti-cancer treatments. If you are called, it should take about 5-10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age: >/= 18 years of age
2. Histologically or cytologically confirmed sarcoma that fall into one of the following categories Patients with low-grade tumors are eligible if there is definite evidence of metastasis or progression (defined as at least a 10% increase in the cumulative sum of the longest diameters within a 3 month period): 1. Adipocytic tumors (Well-differentiated/dedifferentiated liposarcoma, myxoid liposarcoma, pleomorphic liposarcoma) 2. Vascular tumors (leiomyosarcoma, angiosarcoma) 3. Undifferentiated pleomorphic sarcoma 4. Synovial sarcoma 5. Osteosarcoma 6. Other sarcoma histologies
3. Must have received and have progressed, are refractory or intolerant to standard therapy appropriate for the specific sarcoma subtype, if there is a standard therapy for the subtype (i.e. Progressing well-differentiated liposarcoma, clear cell sarcoma etc do not require prior therapy).
4. Subjects must have at least 1 lesion that is measurable by irRECIST a. A previously irradiated lesion can be considered a target lesion if the lesion is well defined, measurable per irRECIST, and has clearly progressed. b. Subjects undergoing fresh tumor biopsies must have additional non-target lesions that can be biopsied at acceptable risk as judged by the investigator or if no other lesion suitable for biopsy, then an irRECIST target lesion used for biopsy must be >/= 2 cm in longest diameter.
5. Subjects must consent to provide archived tumor specimens for correlative biomarker studies. Tumor tissue must be identified and availability confirmed prior to initiation of study therapy. In the setting where archival material is unavailable or unsuitable for use, or there have been multiple intervening therapies subjects must consent and undergo fresh tumor biopsy. A tumor lesion planned for biopsy must not be an irRECIST target lesion unless there are no other lesions suitable for biopsy and lesion used for biopsy is >/= 2 cm in longest diameter.
6. ECOG performance status of 0 or 1
7. Adequate organ function as determined by (lymphocyte count): a. Hematological (without growth factor or transfusion support): i. Absolute neutrophil count >/= 1.5 x 10^9/L (1,500/mm^3) ii. Platelet count >/= 90 × 10^9/L (100,000/mm^3) iii. Hemoglobin >/= 8.0 g/dL within first 2 weeks prior to first dose of investigational product b. Renal: i. Calculated creatinine clearance (CrCl) or 24-hour urine CrCl > 50 mL/min Cockcroft-Gault formula (using actual body weight) will be used to calculate CrCl, except for pts with Osteosarcoma who will be allowed to participate with an estimated creatinine clearance (CrCl) of > 40 mL/min, as calculated by the Cockcroft-Gault equation. c. Hepatic: i. Total bilirubin </= 1.5 × ULN; for subjects with documented/suspected Gilbert's disease, bilirubin </= 3 × ULN ii. AST and ALT </= 2.5 × ULN; for subjects hepatic metastases, ALT and AST </= 5 × ULN
8. Females of childbearing potential who are sexually active with a nonsterilized male partner must use a highly effective method of contraception from the time of screening, and must agree to continue using such precautions for 180 days after the final dose of investigational product.
9. Life expectancy of at least 6 months.
10. Ability to understand the purposes and risks of the study and has signed a written consent form approved by the investigator's IRB/Ethics Committee

Exclusion Criteria:

1. Prior therapy with anti-PD1, anti-PD-L1 or anti-CTLA-4 antibody
2. Active or prior documented autoimmune disease (including inflammatory bowel disease, celiac disease, Wegener syndrome) within the past 2 years. Subjects with childhood atopy or asthma, vitiligo, alopecia, Hashimoto syndrome, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
3. Untreated central nervous system metastatic disease, leptomeningeal disease, or cord compression. Subjects previously treated central nervous system metastases that are radiographically and neurologically stable for at least 6 weeks and do not require corticosteroids (of any dose) for symptomatic management for at least 14 days prior to first dose of MEDI4736 and tremelimumab are permitted to enroll.
4. Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or the follow-up period of an interventional study.
5. Receipt of any conventional or investigational anticancer therapy not otherwise specified above within 28 days or 5 half-lives of the agent prior to the first dose of durvalumab and tremelimumab.
6. Any concurrent chemotherapy, Immunotherapies or biologic or hormonal therapy for cancer treatment. Concurrent use of hormones for non-cancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable. In addition, local treatment (eg, by local surgery or radiotherapy) of isolated lesions for palliative intent is acceptable beyond the first cycle with prior consultation and in agreement with the PI.
7. Unresolved toxicities from prior anticancer therapy, defined as having not resolved to NCI CTCAE v4.03 Grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (eg, hearing loss) after consultation with the study chair.
8. Current or prior use of immunosuppressive medication within 14 days prior to the first dose of MEDI4736 or tremelimumab. The following are exceptions to this criterion: a. Intranasal, inhaled, topical steroids, or local steroid injections (eg, intra-articular injection), b. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent, c. Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication).
9. History of primary immunodeficiency, solid organ transplantation, or previous clinical diagnosis of tuberculosis
10. True positive test results for human immunodeficiency virus (HIV) or hepatitis B or C.
11. Receipt of live, attenuated vaccine within 28 days prior to the first dose of investigational products (NOTE: Subjects, if enrolled, should not receive live vaccine during the study and 180 days after the last dose of investigational products).
12. Major surgery (as defined by the investigator) within 4 weeks or thoracotomy for pulmonary metastases within 2 weeks prior to first dose of treatment or if still recovering from prior surgery. Local surgery of isolated lesions for palliative intent is acceptable.
13. Other invasive malignancy within 2 years except for noninvasive malignancies such as cervical carcinoma in situ, non-melanomatous carcinoma of the skin or ductal carcinoma in situ of the breast that has/have been surgically cured.
14. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from MEDI4736 or tremelimumab, or compromise the ability of the subject to give written informed consent.
15. Any condition that, in the opinion of the investigator or sponsor, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
16. Patients with a history of pneumonitis or interstitial lung disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2016-08-16 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neeta Somaiah, MBBS, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Somaiah N, Conley AP, Parra ER, Lin H, Amini B, Solis Soto L, Salazar R, Barreto C, Chen H, Gite S, Haymaker C, Nassif EF, Bernatchez C, Mitra A, Livingston JA, Ravi V, Araujo DM, Benjamin R, Patel S, Zarzour MA, Sabir S, Lazar AJ, Wang WL, Daw NC, Zhou X, Roland CL, Cooper ZA, Rodriguez-Canales J, Futreal A, Soria JC, Wistuba II, Hwu P. Durvalumab plus tremelimumab in advanced or metastatic soft tissue and bone sarcomas: a single-centre phase 2 trial. Lancet Oncol. 2022 Sep;23(9):1156-1166. doi: 10.1016/S1470-2045(22)00392-8. Epub 2022 Aug 4. PMID 35934010
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Adipocytic Tumors Group: Adipocytic Tumors Group consists of well-diff/de-differentiated, pleomorphic and myxoid LPS.
  Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Durvalumab: Age group ≥ 18: Durvalumab 1500 mg by vein every 4 weeks for 4 cycles. After Week 16, participant may continue to receive durvalumab alone by vein for an additional 32 weeks (8 doses).
  Tremelimumab: Age group ≥ 18: Tremelimumab 75 mg every 4 weeks for 4 cycles.
- Vascular Tumors Group: Vascular Tumors Group consists of leiomyosarcomas, angiosarcomas, epithelioid hemangioendotheliomas, and hemangiopericytomas.
  Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by Durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Durvalumab: Age group ≥ 18: Durvalumab 1500 mg by vein every 4 weeks for 4 cycles. After Week 16, participant may continue to receive durvalumab alone by vein for an additional 32 weeks (8 doses).
  Tremelimumab: Age group ≥ 18: Tremelimumab 75 mg every 4 weeks for 4 cycles.
- Undifferentiated Pleomorphic Sarcoma Group; Synovial Sarcoma Group; Osteosarcoma Group; Other Sarcomas Group; Alveolar Soft-part Sarcoma Group; Chordomas Group: Age group ≥12 and <18: Dosages of study drugs to be determined (TBD).
  Age group ≥ 18: Durvalumab 1500 mg and Tremelimumab 75 mg every 4 weeks for 4 cycles followed by Durvalumab 1500 mg every 4 weeks for up to 8 additional cycles.
  Combination of both agents administered every 4 weeks for a maximum of 4 doses, after which durvalumab continues as a single agent every 4 weeks till progression or unacceptable toxicity for a maximum of 8 additional doses.
  Durvalumab: Age group ≥ 18: Durvalumab 1500 mg by vein every 4 weeks for 4 cycles. After Week 16, participant may continue to receive durvalumab alone by vein for an additional 32 weeks (8 doses).
  Tremelimumab: Age group ≥ 18: Tremelimumab 75 mg every 4 weeks for 4 cycles.
Period: Overall Study
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group
Started | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5
Completed | 2 | 1 | 1 | 1 | 2 | 1 | 6 | 4
Not Completed | 4 | 9 | 4 | 4 | 3 | 10 | 4 | 1
Not completed — Disease Progression | 3 | 7 | 2 | 4 | 3 | 9 | 3 | 1
Not completed — Adverse Event | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group | Total
Number analyzed (Participants) | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.24 (8.39) | 53.68 (13.14) | 55.18 (16.32) | 35.97 (9.13) | 45.84 (17.42) | 44.49 (15.95) | 34.09 (9.88) | 61.76 (6.97) | 48.18 (15.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 1 | 3 | 2 | 4 | 6 | 1 | 26
  Male | 5 | 2 | 4 | 2 | 3 | 7 | 4 | 4 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 1 | 5
  Not Hispanic or Latino | 6 | 9 | 5 | 5 | 4 | 11 | 8 | 4 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 4
  White | 6 | 9 | 5 | 4 | 3 | 10 | 4 | 4 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5 | 57

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20%increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 12 weeks
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group
Number analyzed (Participants) | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5
proportion of participants | 0.17 [0.01 to 0.52] | 0.3 [0.07 to 0.58] | 0.4 [0.05 to 0.75] | 0.8 [0.2 to 0.97] | 0.2 [0.01 to 0.58] | 0.45 [0.17 to 0.71] | 0.9 [0.47 to 0.99] | 0.8 [0.2 to 0.97]

2. Secondary Outcome: Tumor Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR),Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 8 weeks, confirmatory scan at least 4 wks or later
Measure: Count of Participants; unit: Participants
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group
Number analyzed (Participants) | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5
Participants
  Best Response irRC - N/A | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Best Response irRC - PD | 3 | 7 | 2 | 1 | 3 | 5 | 1 | 1
  Best Response irRC - PR | 0 | 1 | 1 | 0 | 0 | 0 | 5 | 1
  Best Response irRC - SD | 3 | 1 | 1 | 2 | 1 | 3 | 4 | 3
  Best Response irRC - uPD | 0 | 1 | 1 | 2 | 0 | 3 | 0 | 0
  Best Response iRecist - N/A | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Best Response iRecist - PD | 3 | 7 | 2 | 0 | 3 | 5 | 1 | 1
  Best Response iRecist - PR | 0 | 1 | 1 | 0 | 0 | 0 | 4 | 1
  Best Response iRecist - SD | 3 | 1 | 1 | 3 | 1 | 3 | 5 | 3
  Best Response iRecist - uPD | 0 | 1 | 1 | 2 | 0 | 3 | 0 | 0

3. Secondary Outcome: Overall Survival (OS)
Description: OS defined as the time from treatment onset to death. OS estimated using the Kaplan-Meier method.
Time Frame: 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group
Number analyzed (Participants) | 6 | 10 | 5 | 5 | 5 | 11 | 10 | 5
months | 10.99 [2.1 to NA] — Not reached. Insufficient number participants with events. | 16.41 [4.47 to 24.87] | 4.99 [1.51 to 30.85] | 32.79 [7.46 to NA] — Not reached. Insufficient number participants with events. | 7.72 [1.38 to 21.59] | 13.31 [3.84 to 25.33] | NA [14.32 to NA] — Not reached. Insufficient number participants with events. | NA [NA to NA] — Not reached. Insufficient number participants with events.

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Adipocytic Tumors Group | Vascular Tumors Group | Undifferentiated Pleomorphic Sarcoma Group | Synovial Sarcoma Group | Osteosarcoma Group | Other Sarcomas Group | Alveolar Soft-part Sarcoma Group | Chordomas Group
All-Cause Mortality (participants affected / at risk) | 4/6 | 8/10 | 5/5 | 4/5 | 5/5 | 10/11 | 2/10 | 0/5
Serious Adverse Events (participants affected / at risk) | 5/6 | 7/10 | 4/5 | 0/5 | 4/5 | 8/11 | 6/10 | 1/5
Other Adverse Events (participants affected / at risk) | 2/6 | 3/10 | 2/5 | 1/5 | 2/5 | 5/11 | 4/10 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adipocytic Tumors Group (N=6) | Vascular Tumors Group (N=10) | Undifferentiated Pleomorphic Sarcoma Group (N=5) | Synovial Sarcoma Group (N=5) | Osteosarcoma Group (N=5) | Other Sarcomas Group (N=11) | Alveolar Soft-part Sarcoma Group (N=10) | Chordomas Group (N=5)
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Autoimmune disorder (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fever (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Unintended pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flu (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Disease Progression (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute renal insufficiency (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Remove tumor (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
chest (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal obstruction (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasms benign, malignant and unspecified (including cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
fracture right femur (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adipocytic Tumors Group (N=6) | Vascular Tumors Group (N=10) | Undifferentiated Pleomorphic Sarcoma Group (N=5) | Synovial Sarcoma Group (N=5) | Osteosarcoma Group (N=5) | Other Sarcomas Group (N=11) | Alveolar Soft-part Sarcoma Group (N=10) | Chordomas Group (N=5)
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Serum amylase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Autoimmune disorder (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Thrush (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1 | 1 | 1 | 3 | 3 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Thyroiditis (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Endocrine disorders - Other, specify (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 1 | 2 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 0 | 4 | 2
Rash (left shoulder) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Left Leg) (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 1 | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Fever (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Flu like symptoms (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash lower back (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-10): https://cdn.clinicaltrials.gov/large-docs/95/NCT02815995/Prot_SAP_000.pdf